CLINICAL TRIAL: NCT00342550
Title: Cervical Volume by Three-Dimensional Ultrasound as a Predictor of Preterm Delivery
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999998016; OH98-CH-N016
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Pregnancy; Preterm Birth; Cervical Length Measurement
Keywords: Pregnancy; Preterm Birth; Pregnancy Complications; Natural History
MeSH Terms: conditions — Premature Birth; Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Pregnant Women: Pregnant women aged 15 and older between 20 and 35 weeks with singleton gestation

SUMMARY:
Preterm labor is a leading cause of perinatal morbidity and mortality. Several investigators have reported that ultrasound evaluation of the cervix can predict the risk of preterm delivery. Three-dimensional ultrasound may provide additional information about how to best counsel parents about the chances of premature birth. This technology has the capability for accurate volume measurements of irregular structures that is superior to conventional ultrasound. Therefore, it is possible that three-dimensional ultrasound methods may better characterize cervical changes and the risk for preterm delivery.

Our protocol will attempt to identify prognostic indicators of adverse pregnancy outcome by three-dimensional ultrasound. A maximum of 680 pregnant women with the diagnosis of preterm labor will be prospectively studied to characterize cervical morphology and volume as predictors of preterm delivery risk. These results will be correlated with placental pathology and pregnancy outcome. We will also compare the performance of conventional two-dimensional endovaginal ultrasound with three-dimensional ultrasound findings. This information is expected to improve our understanding about the nature and timing of cervical volume changes in relation to pregnancy outcome.

DETAILED DESCRIPTION:
Preterm labor is a leading cause of perinatal morbidity and mortality. Several investigators have reported that ultrasound evaluation of the cervix can predict the risk of preterm delivery. Three-dimensional ultrasound may provide additional information about how to best counsel parents about the chances of premature birth. This technology has the capability for accurate volume measurements of irregular structures that is superior to conventional ultrasound. Therefore, it is possible that three-dimensional ultrasound methods may better characterize cervical changes and the risk for preterm delivery.

Our protocol will attempt to identify prognostic indicators of adverse pregnancy outcome by three-dimensional ultrasound. A maximum of 680 pregnant women with the diagnosis of preterm labor will be prospectively studied to characterize cervical morphology and volume as predictors of preterm delivery risk. These results will be correlated with maternal and fetal biological markers, placental pathology and pregnancy outcome. We will also compare the performance of conventional two-dimensional endovaginal ultrasound with three-dimensional ultrasound findings. This information is expected to improve our understanding about the nature and timing of cervical volume changes in relation to pregnancy outcome.

ELIGIBILITY:
* INCLUSION CRITERIA - PRETERM LABOR AND INTACT MEMBRANES:

  1. Singleton gestation;
  2. Estimated gestational age between 20 and 35 weeks gestation;

  3 Intact membranes;

  4. Signed informed consent for voluntary participation and serial endovaginal scans.

EXCLUSION CRITERIA - PRETERM LABOR AND INTACT MEMBRANES:

1. Absent fetal cardiac activity;
2. Desire not to have vaginal ultrasound scans.

INCLUSION CRITERIA - PATIENTS AT RISK FOR PRETERM DELIVERY:

1. Estimated gestational age between 16 and < 24 weeks gestation;
2. Planned cerclage placement due to increased preterm labor risk (i.e., short cervix or dilated cervix);
3. Intact membranes;
4. Signed informed consent for voluntary participation and serial endovaginal scans.

EXCLUSION CRITERIA - PATIENTS AT RISK FOR PRETERM DELIVERY:

1. Absent fetal cardiac activity;
2. Desire not to have vaginal ultrasound scans.

INCLUSION CRITERIA - PATIENTS IN SPONTANEOUS LABOR AT TERM:

1. Term gestation (greater than 37 weeks);
2. Intact membranes;
3. Cervical dilatation less than 2 cm;
4. Signed informed consent for voluntary participation and serial endovaginal scans.

EXCLUSION CRITERIA - PATIENTS IN SPONTANEOUS LABOR AT TERM:

1. Absent fetal cardiac activity;
2. Desire not to have vaginal ultrasound scans.

INCLUSION CRITERIA - PATIENTS UNDERGOING ELECTIVE INDUCTION OF LABOR:

1. Term gestation (greater than 37 weeks);
2. Intact membranes;
3. Signed informed consent for voluntary participation and serial endovaginal scans.

EXCLUSION CRITERIA - PATIENTS UNDERGOING ELECTIVE INDUCTION OF LABOR:

1. Absent fetal cardiac activity;
2. Desire not to have vaginal ultrasound scans.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women attending Hutzel Women's clinic at Detroit Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 648 (Actual)
Dates: Start 1998-03-11 (Actual); Primary Completion 2008-05-01 (Actual); Study Completion 2008-05-01 (Actual)

PRIMARY OUTCOMES:
Document cervical volume and funneling changes in women with preterm labor. Determine the relationship between cervical volume and funneling changes to the risk of preterm delivery. | Ongoing
  Data analysis is ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Romero, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- Hutzel Women's Hospital, Detroit, Michigan, United States

REFERENCES:
- [Background] Ayers JW, DeGrood RM, Compton AA, Barclay M, Ansbacher R. Sonographic evaluation of cervical length in pregnancy: diagnosis and management of preterm cervical effacement in patients at risk for premature delivery. Obstet Gynecol. 1988 Jun;71(6 Pt 1):939-44. PMID 3285274